CLINICAL TRIAL: NCT06991049
Title: Early Versus Late Endoscopic Temporary Stenting for Management of Refractory Benign Esophageal Strictures
Brief Title: Early Versus Late Endoscopic Stenting for Refractory Benign Esophageal Strictures
Acronym: RBES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Kulwinder Dua, MD, Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00054233
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Refractory Benign Esophageal Strictures
Keywords: Refractory Benign Esophageal Strictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Late-stent approach (Active Comparator): Repeated dilations at weekly intervals, and based on the response, the intervals between dilations are adjusted, and if still no response, place a removable FCSEMS (18 mm diameter). The stent will be removed in 2 weeks followed again by weekly dilations till less than one dilation is needed every 3 months to maintain a luminal diameter of 14 mm or more.
  Interventions: Device: Fully covered self-expandable metal esophageal stent
- Early-stent approach (Active Comparator): Removable FCSEMS (18 mm diameter) placed on index endoscopy and removed after 2 weeks followed by weekly dilations till less than one dilation is needed every 3 months to maintain a luminal diameter of 14 mm or more.
  Interventions: Device: Fully covered self-expandable metal esophageal stent

INTERVENTIONS:
Device: Fully covered self-expandable metal esophageal stent — Esophageal stent placement for patients with benign esophageal strictures not responding to endoscopic dilations.

SUMMARY:
This project is being done to compare two current treatment clinical options for management of RBES: 1) Frequent dilations followed by temporary esophageal stent placement if dilations fail, or 2) Early stent placement followed by dilations

DETAILED DESCRIPTION:
This study aims to explore the safety and effectiveness of two clinical treatment approaches used to manage RBES patients-Temporary early-stent placement versus late stenting.

For normal swallowing, the esophagus (food pipe) lumen should be equal to or more than 14 mm in diameter. In those with stricture (narrowing) of the esophagus from benign causes, initial endoscopic management is serial sessions of dilation (stretching) to achieve and maintain a diameter of ≥14mm. Many strictures may not respond to this approach (refractory). Esophageal stents (18 mm - 23 mm diameter) temporarily placed for 2 weeks using an endoscope are also used dilate and remold the stricture. While in place, patients can swallow. This can save the patient from undergoing repeated dilations. Stents can be placed either late in the process of management after several traditional dilations have failed or early in the management to rapidly achieve a diameter of ≥14 mm and then continuing traditional dilations.

Although either of above two approaches can be used for the clinical management of RBES, in this study the investigators plan to randomly assign patients to start with one of the two approaches and compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed and written consent.
* Able to keep follow up appointments as per protocol (minimum 2 years).
* Biopsy proven benign esophageal stricture.
* Dysphagia (grade 2 and above).
* Fit to undergo upper GI endoscopy.
* Documented esophageal stricture with a luminal diameter <14 mm at index endoscopy.

Exclusion Criteria:

* Minimal dysphagia (grade 0-1)
* Neuromuscular dysphagia (such as achalasia, oro-pharyngeal dysphagia post-stroke, crico-pharyngeal bar, Zenker diverticulum etc.)
* Pregnant or planning to be pregnant during the study period.
* Malignant or indeterminate esophageal stricture.
* Actively receiving radiation therapy.
* Persistent associated active esophagitis that has not yet healed.
* Esophageal strictures associated with fistula/leaks/current or prior perforation.
* Eosinophilic esophagitis.
* Associated esophageal varices.
* No other malignancy limiting life expectancy.
* Patients in whom placing esophageal stents is not possible/contraindicated (such as high cervical esophageal strictures, active bleeding, metal allergy, tortuous esophagus, pseudodiverticulum with stricture).
* Previous esophageal stent tried over 2 months ago
* Significant comorbidities making patient high risk for upper GI endoscopy.
* Unable to give informed consent.
* Cannot keep follow up appointments as per protocol.
* Procedures and stents not covered by patient's insurance.
* Patients who, after comprehensive discussion and explanation of both the early-stent and late-stent approaches, choose to proceed with a specific approach and decline participation in randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-03-21 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to achieve esophageal luminal diameter to ≥14 mm | From enrollment to follow up, up to 2 years
  The duration required to achieve and maintain an esophageal diameter of ≥14 mm using the two techniques.

SECONDARY OUTCOMES:
Adverse event rate | From enrollment to follow up, up to 2 years
Recurrence rate of esophageal stricture | From enrollment to follow up, up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No